CLINICAL TRIAL: NCT00500344
Title: CAPTAIN: Choroidal Neovascularization Assessment by Pattern Electroretinography After Ranibizumab in Naive Age-related Macular Degeneration Patients
Brief Title: CAPTAIN:Choroidal Neovascularization Assessment by Pattern Electroretinography
Acronym: CAPTAIN
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Rajendra S. Apte, Rajendra S. Apte MD, PHD, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FVF4184S
Record Dates: First submitted 2007-07-10; First posted 2007-07-12 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Age-related Macular Degeneration
Keywords: Age-related Macular Degeneration; Choroidal Neovascularization; Electroretinography; Retinal Function
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other)
  Interventions: Drug: Lucentis (ranibizumab)

INTERVENTIONS:
Drug: Lucentis (ranibizumab) — intravitreal injection

SUMMARY:
CNV from AMD is the leading cause of blindness in people over 50 in North America. The hypothesis is to determine if there is an improvement in retinal function determined by ERG following treatment with ranibizumab for AMD

DETAILED DESCRIPTION:
1. Background 1.1 Pathophysiology Age-related macular degeneration (AMD) is a progressive disease that causes irreversible visual impairment and blindness in nearly 50 million people globally 1. 2. Current estimates of patients affected with AMD are higher than those affected by Alzheimer's disease 1.3 Although geographic atrophy and neovascularization represent the advanced forms of AMD, neovascular AMD is the more aggressive form and accounts for almost 90% of blindness from this disease. It is characterized by choroidal neovascularization (CNV) which is the development of abnormal blood vessels underneath the retina. Current treatments such as photodynamic therapy (PDT) and intravitreal pegaptanib are designed to limit further visual loss, but these are only marginally effective 4-6.

   1.2 Treatment of on-label naive AMD patients Recent randomized clinical trials (Marina, Anchor) have conclusively demonstrated that continued intravitreal therapy with ranibizumab in patients with subfoveal CNV from AMD leads to stabilization of vision in over 90% of patients and improvement in vision in at least a third of the patients and has led to the approval of ranibizumab (0.5 mg) for the treatment of neovascular AMD. Naive patients will be used in this study to determine if an improvement by ERG can be determined in those without prior therapy.

   1.3 Electroretinography(ERG) Effects Of Ranibizumab Therapy AMD trials are typically designed to address visual acuity outcomes but not designed to evaluate retinal function outcomes. Global and macular retinal indices as measured by electroretinography (ERG) are key indicators of retinal health which have largely been ignored in clinical trials.

   1.4 Non-Clinical Experience With Ranibizumab 1.4.1 Nonclinical Pharmacokinetics The pharmacokinetics of ranibizumab have been investigated in rabbits and cynomolgus monkeys following intravitreal and intravenous administration. In both species, following intravitreal administration, ranibizumab was cleared from the vitreous humor with a half life of 2-3 days. Following single intravitreal administration to cynomolgus monkeys, retinal concentrations of ranibizumab were approximately one third of vitreous concentrations and declined in parallel with vitreous concentrations. In humans, the intravitreal half-life of ranibizumab is estimated to be 7-8 days. Repeated intravitreal injections of ranibizumab can lead to detectable antibodies in serum in rabbits and cynomolgus monkeys.

   1.4.2 Nonclinical Toxicology A series of nonclinical studies of ranibizumab administered by intravitreal injection to cynomolgus monkeys have been performed (details regarding study design and results can be found in the Investigator Brochure).

   1.4.3 Stability Studies The stability of ranibizumab alone and in combination with verteporfin was assessed in vitro. The combination of ranibizumab and verteporfin in a 5% dextrose solution at concentrations of 500 mg/mL and 1.4 mg/mL, respectively, resulted in ranibizumab degradation and a decrease in ranibizumab capacity to bind VEGF. The ranibizumab degradation products have not been fully characterized. Although it is currently unknown if such degradation also occurs in vivo, sequential administration of verteporfin followed by ranibizumab with an intervening washout period will decrease the likelihood of loss of ranibizumab activity and degradation.

   1.5 Clinical Experience With Ranibizumab Ranibizumab has been or is being clinically evaluated in nine studies (additional details regarding study design and results can be found in the Investigator Brochure).

   The first clinical trial with ranibizumab, Study FVF1770g was a Phase Ia study of the molecule given as a single intravitreal injection to subjects with neovascular AMD. The goals of the study were to investigate safety and tolerability and to define the maximally tolerated dose (MTD). The single intravitreal MTD was determined to be 0.5 mg (limited by ocular inflammation).

   The Phase I/II study FVF2128g was the first clinical trial of multiple-dose regimens of intravitreally administered ranibizumab. Sixty-four subjects were enrolled in the study. Data show that ranibizumab was safe and potentially efficacious in subjects with subfoveal choroidal neovascularization due to AMD.

   Study FVF2425g was a Phase I, open-label, randomized study of three escalating multiple dose regimens of intravitreally administered ranibizumab. Data show that doses of ranibizumab up to 2 mg could be safely given as part of an escalating dose regimen to subjects with subfoveal choroidal neovascularization due to AMD.

   Study FVF2428g was a Phase I/II, single masked, multicenter study of the safety, tolerability, and efficacy of multiple dose intravitreal injections of ranibizumab in combination with verteporfin PDT in subjects with neovascular AMD. Data show that the combination of ranibizumab and verteporfin PDT had a good safety profile in the study population, and the efficacy of ranibizumab and verteporfin PDT was better than that of verteporfin PDT alone.

   Preliminary findings from Study FVF2428g suggest that administration of ranibizumab injections 7 days (plus/minus 2 days) after treatment with verteporfin PDT in the same eye may result in a decrease in visual acuity of 30 letters due to temporary intraocular inflammation (uveitis).

   Study FVF2508g is an ongoing Phase I extension study designed to assess the safety and tolerability of multiple-dose intravitreal injections of ranibizumab administered monthly in subjects who have completed the treatment phase of a Genentech-sponsored Phase I study.

   Study FVF2587g is an ongoing Phase III active treatment-controlled study designed to assess the efficacy and safety of intravitreal administered ranibizumab compared with verteporfin in subjects with angiographically determined, predominantly classic subfoveal neovascular AMD.

   Study FVF2598g was an ongoing Phase III study designed to assess the efficacy and safety of intravitreal injections of ranibizumab administered monthly compared with sham injections administered monthly in subjects with angiographically determined, minimally classic or occult subfoveal neovascular AMD. Data show that ranibizumab was safe and efficacious in subjects with subfoveal CNV due to AMD.

   Study FVF3192g is an ongoing Phase IIIb study designed to assess the efficacy and safety of intravitreal injections of ranibizumab administered as three monthly injections followed by quarterly injections for a total duration of 24 months, in subjects with angiographically determined subfoveal neovascular AMD with or without classic CNV.

   Study 3426g is an ongoing open-label extension study designed to assess the safety and tolerability of intravitreal injections of ranibizumab in subjects who have completed the treatment phase of a Genentech-sponsored ranibizumab study.

   Study 3689g is an ongoing Phase IIIb, 1 year multicenter study of the safety and tolerability of intravitreally administered ranibizumab at two different doses (0.3mg and 0.5mg) to subjects with active subfoveal CNV secondary to AMD, administered once a month for 3 months and thereafter as needed, based on criteria-based re-treatment options.
2. Objectives

   2.1 Primary Objective To determine if there is an improvement in retinal function determined by the pattern and full-field ERG following treatment with ranibizumab for AMD

   2.2 Secondary Objectives To determine if there is a correlation between improvement in visual acuity and retinal function as determined by the ERG Visual acuity at 6 months
3. Study Design 3.1 Description Of The Study This is an open-label, Phase I single arm study of intravitreally administered ranibizumab in on-label treatment naive patients following by an assessment of retinal function using the ERG.

Consented, enrolled subjects will receive monthly open-label intravitreal injections of 0.5 mg ranibizumab administered every month for 6 months. ERG will be performed at baseline, 1 month, 3 months and 6 months.

Electroretinograms will be recorded using DTL fiber electrodes moistened with carboxymethyl-cellulose sodium 1% lying in the inferior fornix of each eye. Each DTL fiber will be laid along the top of the lower eyelids so that it contacts the inferior cornea. Fibers will be anchored with small adhesive pads near the inner and outer canthi. A reference electrode will be applied with adhesive paste lateral to the outer canthi. An adhesive electrode placed on the forehead will serve as the ground. Prior to pupil dilation, PERG responses will be recorded, including P50 (derived from macular photoreceptors) and N95 (post-photoreceptor, including optic nerve), in response to an alternating checkerboard pattern. Pupils will then be dilated with tropicamide 1% and phenylephrine hydrochloride 2.5% for the full-field ERG and PhNR recordings. The patient will be dark-adapted for 30 minutes. For full-field recordings, stimuli will be brief white flashes presented by a Ganzfeld integrating sphere. Responses to dim and bright flashes will be recorded under scotopic conditions, and a- and b-wave amplitudes will be noted. Patients will then be light adapted for ten minutes. Responses to bright flash and 30 Hz flicker responses will then be recorded under photopic conditions. A- and b-wave amplitudes and implicit times will be noted. Finally, the photopic negative response (PhNR) will be recorded with a red flash on a blue background.

3.2 Rationale For Study Design Per the package insert, naive AMD patients will receive monthly injections of Lucentis as part of their usual care.

3.3 Outcome Measures 3.3.1 Primary Outcome Measures Percent of patients with Improvement in ERG from baseline to 6 months based on international standards (determined by expert reader).

3.3.2 Secondary Outcome Measures

Percent of patients with Improvement in ERG from baseline to 3 months based on international standards (determined by expert reader) Correlation between change in PERG and mean change in VA at 6 months Mean change in VA from baseline to 3 months and 6 months.

3.4 Safety Plan There are no safety issues associated with the ERG. All safety monitoring will be as in standard care with the use of on-label ranibizumab. ERG testing is non-invasive.

3.5 Compliance With Laws And Regulations This study will be conducted in accordance with current U.S. Food and Drug Administration (FDA) Good Clinical Practices (GCPs), and local ethical and legal requirements.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age ≥ 50 years
* Treatment naive AMD patients that are determined to be candidates for ranibizumab
* Visual acuity 20/40 to 20/320

Exclusion Criteria:

* Pregnancy
* Prior enrollment in the study
* Previous therapy for AMD or other retinal diseases which may be used in the treatment of AMD
* Any other condition that the investigator believes would pose a significant hazard to the subject if on-label ranibizumab were prescribed
* Any condition that would interfere with the ERG recording (such as media opacities including lens or corneal opacity)
* Concurrent eye disease in the study eye that could compromise visual acuity (such as diabetic retinopathy, advanced glaucoma)
* Any condition causing the patient to have a significant tremor that would interfere with the patient's ability to remain still during the ERG (such as Parkinson's disease)
* Participation in another simultaneous medical investigation or trial

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To determine if there is an improvement in retinal function determined by the ERG following treatment with ranibizumab | 6 months

SECONDARY OUTCOMES:
To determine if there is an improvement in visual acuity and retinal function as determined by ERG | 6 months
Correlation between change in PERG and mean change in VA at 6 months | 6 months
Mean change in VA from baseline to 0 months and 6 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Rajendra S. Apte, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

REFERENCES:
- [Background] Klein R, Peto T, Bird A, Vannewkirk MR. The epidemiology of age-related macular degeneration. Am J Ophthalmol. 2004 Mar;137(3):486-95. doi: 10.1016/j.ajo.2003.11.069. PMID 15013873
- [Background] van Leeuwen R, Klaver CC, Vingerling JR, Hofman A, de Jong PT. Epidemiology of age-related maculopathy: a review. Eur J Epidemiol. 2003;18(9):845-54. doi: 10.1023/a:1025643303914. PMID 14561043
- [Derived] Sheybani A, Brantley MA Jr, Apte RS. Pattern electroretinography in age-related macular degeneration. Arch Ophthalmol. 2011 May;129(5):580-4. doi: 10.1001/archophthalmol.2011.83. PMID 21555610